CLINICAL TRIAL: NCT00759096
Title: Clinical Assessment of Visual Function With the Acrysof ReSTOR Multifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-06-03
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-02-10 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2010-01

CONDITIONS: Visual Acuity
Keywords: bilateral implantation; ReSTOR Aspheric IOL; uniocular unaided distance; binocular unaided distance; intermediate visual acuity; near visual acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acrysof ReSTOR IOL (Experimental): AcrySof ReSTOR Intraocular lens (IOL) implanted
  Interventions: Device: RESTOR IOL Model SA60D3

INTERVENTIONS:
Device: RESTOR IOL Model SA60D3 — Implanted into the study eye following cataract extraction surgery

SUMMARY:
The purpose of this study is to assess uniocular and binocular unaided distance, intermediate, and near VA; contrast sensitivity, accommodation amplitude, stereopsis, glare testing, ocular aberrations and the clinical satisfaction assessment after bilateral implant of the Restor IOL.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of either gender or any race
* Potential post-op VA 20/20
* Pre-op astigmatism ≤ 1.0D
* Able to sign the informed consent
* Able to complete all required postoperative visits
* Planned cataract removal by phaco
* Clear intraocular media other than cataract

Exclusion Criteria:

* Signs of capsular tear, significant anterior chamber hyphema, or zonular rupture
* Any corneal pathology and previous corneal refractive surgery
* Patients with unrealistic expectations in anticipated post-op VA
* Happy to wear glasses
* Occupational night driver

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients with bilateral cataract were implanted with ReSTOR lens and followed up for 6-month after the 2nd eye implantation
Pre-assignment Details: Open-label, single arm and nonrandomized
Groups:
- AcrySof ReSTOR IOL: Acrysof ReSTOR Intraocular Lens (IOL)
Period: Overall Study
Arm/Group | AcrySof ReSTOR IOL
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AcrySof ReSTOR IOL
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Near Uncorrected Visual Acuity(UCVA
Description: Near uncorrected visual acuity(UCVA) measured in logMAR. LogMAR is the logarithm of the minimum angle of resolution and is used to measure visual acuity.
Time Frame: 6 months after surgery of 2nd eye
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof ReSTOR IOL
Number analyzed (Participants) | 30
logMAR | 0.5 (0.12)

2. Secondary Outcome: Contrast Sensitivity
Time Frame: 6 months after sugery of the 2nd eye
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | AcrySof ReSTOR IOL
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No